CLINICAL TRIAL: NCT03933722
Title: Comparison of Noninvasive Blood Pressure Monitoring With Invasive Arterial Pressure Monitoring in Patients With Septic Shock
Brief Title: Caretaker vs. Blood Pressure Monitoring With Invasive Arterial Pressure Monitoring in Patients With Septic Shock
Status: Active, not recruiting | Type: Observational
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 18-180EX
Record Dates: First submitted 2019-04-18; First posted 2019-05-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Caretaker: Comparing blood pressure obtained using routine blood pressure sphygmomanometer to a non-invasive device that continuously monitors central blood pressure (CareTaker).
  Interventions: Device: Caretaker

INTERVENTIONS:
Device: Caretaker — Application of Caretaker device to subjects that have septic shock and that have an invasive arterial pressure monitor placed.

SUMMARY:
Caretaker vs. Blood Pressure Monitoring With Invasive Arterial Pressure Monitoring in Patients With Septic Shock

DETAILED DESCRIPTION:
The aim of this study is to compare blood pressure obtained using routine blood pressure sphygmomanometer, in patients with invasive arterial pressure monitoring that have septic shock, to a non-invasive device that continuously monitors central blood pressure (CareTaker).

ELIGIBILITY:
Inclusion Criteria:

* Admitted with septic shock, with or without vasopressor support needed.
* Greater than or equal to 18 years of age.
* Have an arterial catheter already in place.

Exclusion Criteria:

* No arterial catheter in place.
* Contraindication to the application of the Caretaker device due to pre-existing finger injury.
* Patients in whom use of a BP cuff is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ages > 18 who have septic shock and have an arterial line monitor in place.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-02-05 (Estimated)

PRIMARY OUTCOMES:
Comparing blood pressure measurements by the Caretaker device to blood pressure measurements made with an intra-arterial pressure catheter. | 20 minutes
  The primary outcome measure will be the average difference in systolic and diastolic blood pressure measurements between the investigational device (Caretaker) and the reference (intra-arterial catheter pressure) in subjects that have septic shock. In line with blood pressure validation guidelines, we will obtain multiple investigational-reference measurement pairs in each subject (20 minutes total) and will average the difference over all pairs from all subjects.

SECONDARY OUTCOMES:
Comparing blood pressure measurements by the Caretaker device to blood pressure measurements made with an upper arm cuff. | 20 minutes
  Secondary outcome measure will be the average difference in systolic and diastolic blood pressure measurements between the investigational device (Caretaker) and a brachial cuff in subjects that have septic shock. In line with blood pressure validation guidelines, we will obtain multiple investigational-reference measurement pairs in each subject (4 pairs over 20 minutes) and will average the difference over all pairs from all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Gratz, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States